CLINICAL TRIAL: NCT02932033
Title: Randomized Control Trial Comparing Tack Versus Histoacryl Mesh Fixation After Endoscopic TEP (Total Extraperitoneal) Repair for Groin Hernias
Brief Title: Trial Comparing Tack Versus Histoacryl Mesh Fixation After Endoscopic TEP(Total Extraperitoneal) Repair for Bilateral Inguinal Hernia
Acronym: TEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Yao-Chou Tsai, Principle investigator, Principal investigator, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 05-X18-072
Record Dates: First submitted 2016-06-28; First posted 2016-10-13 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tack fixation (Active Comparator): consecutive patients with bilateral inguinal hernias will be recruited for TEP repair. Mesh fixation methods with spiral tack is randomly assigned to one side, then comparative fixation method to the contralateral side. In group of active comparator, after randomization, the target inguinal hernia side of the patient has the mesh fixed with titanium spiral tacks.
  Interventions: Procedure: Tack fixation of mesh
- Synthetic glue fixation (Experimental): The same patient, his contralateral side of inguinal hernia, has the mesh fixed with synthetic glue.
  Interventions: Procedure: Synthetic glue fixation

INTERVENTIONS:
Procedure: Tack fixation of mesh — hernia mesh is fixed with synthetic glue (Histoacryl) (experimental) or spiral titanium tacks (active comparator) according to the result of randomization
  Arms: Tack fixation
Procedure: Synthetic glue fixation — hernia mesh is fixed with synthetic glue (Histoacryl) (experimental) according to the result of randomization
  Arms: Synthetic glue fixation

SUMMARY:
This prospective randomized trial is performed to analyze the post-operative pain (acute and chronic) after endoscopic TEP repair after bilateral inguinal hernia repair.

DETAILED DESCRIPTION:
consecutive patients with bilateral inguinal hernias will be recruited for TEP repair. Mesh fixation methods spiral tacks glue is randomly assigned to one side to the groin and Histoacryl synthetic glue to the other side. Patients will be followed up regularly for up to 6 months by an independent clinical nurse was blinded to the mesh fixation assignment. The patients are also blinded to the the mesh fixation assignment. The post operative pain score, peri-operative complication, and recurrences will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients present with clinical bilateral inguinal hernias And feasible for general anesthesia

Exclusion Criteria:

* Patient preference for either fixation technique, refusal to participate, previous major lower abdominal surgery, concomitant surgical procedures other than hernia repair, and history of allergy to Histoacryl.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
acute post-operative pain with VAS | 6 hours after OP

SECONDARY OUTCOMES:
Chronic pain VAS pain scale | 6 months after OP
Questionnaire of complications | 6 months after OP

CONTACTS AND LOCATIONS:
Locations (1):
- Buddhist Tzu Chi General Hospital, Taipei branch, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No